CLINICAL TRIAL: NCT05867706
Title: The Psychobiological Adjustment to Bereavement Among Cancer Caregivers
Brief Title: Caregiver Stress and Bereavement
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: University of Salzburg (Other); University of California (Other)
Responsible Party: Sponsor
Other Study IDs: KLS-5643-08-2022
Record Dates: First submitted 2023-03-09; First posted 2023-05-22 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Caregiver Burden; Bereavement; Cancer
Keywords: caregiver; bereavement; stress; biomarkers; cancer; palliative care
MeSH Terms: conditions — Caregiver Burden; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nail clip blood serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The death of a spouse is considered one of the most stressful and impactful life events and is associated with increased morbidity and premature mortality. Early identification of individuals who are most at risk for poor health outcomes following bereavement is an important aim of precision medicine and disease prevention initiatives. A better understanding of caregiver burden and bereavement-related distress and its implication for health is a clinically-relevant step toward the development of treatments that improve health outcomes in bereaved spouses. This study aims to map profiles of individual differences in short- and long-term adjustment to loss, according to psychological (e.g., depression, stress, grief severity) and biological markers (e.g., inflammation, cortisol) over time.

DETAILED DESCRIPTION:
The loss of a spouse is a highly impactful life event that places individuals at risk for mental and physical health problems. Particularly in the immediate weeks and months after the loss, bereavement is associated with a significantly increased risk of multimorbidity and mortality, including elevated inflammation, cardiovascular diseases and some cancers. Grief is a typical reaction to the loss of a significant person and is characterized by symptoms of intense distress, anxiety, yearning, longing, and sadness, all of which generally subside over time. There is considerable variability in how people respond to bereavement. Although the vast majority of bereaved individuals show resilience against loss and adjust adequately without professional psychological support, 10% - 20% of bereaved individuals develop intense and prolonged grief reactions.

The field of psychoneuroimmunology has contributed considerably to our understanding of the effect of stress on the psyche, as well as on the nervous, immune, and endocrine systems. Stressful life events, and the negative emotions they provoke, can induce low-grade inflammation through several autonomic, neuroendocrine, and neuroimmune pathways, which in turn suppress the effectiveness of the immune system, and thereby, increase vulnerability to physical and mental health problems across a person's lifespan. Bereavement is a highly-stressful event, which triggers biological responses via several autonomic, endocrine, and inflammatory mechanisms. Growing evidence suggests that the health consequences of caregiving for terminally-ill patients and bereavement after the loss of a spouse are associated with a wide spectrum of neuroendocrine factors and immunologic and inflammatory markers. Low-grade systemic inflammation, as reflected by elevated concentrations of cytokines (e.g., C-reactive protein, CRP; interleukin 6, IL-6; tumor necrosis factor alpha, TNF-a) is a robust risk factor for the onset of many diseases, including major depression, cardiovascular disease, and stroke.

The caregivers' burden and needs are often not a hospital's priority and overlooked. Yet, the health consequences of caring for a terminally-ill spouse, as well as the need for follow-up care programs for caregivers of a deceased spouse are not well understood. Acknowledging that bereavement-related changes in immune function could account considerably for an increased risk of morbidity and mortality in bereaved individuals, the identification of biobehavioral mechanisms that can be modified or targeted early is an important and clinically-relevant step toward the development of treatments that improve health outcomes in bereaved individuals.

The proposed study is based on the Social Signal Transduction Theory of Depression (Slavich et al.), which suggests that early life stress exposure can shape an individual's neuro-inflammatory sensitivity to stress to later- occurring threats or acute adverse life events, and thereby increase their vulnerability to physical and mental health problems across the lifespan.

The study's aims are two-fold: 1) to map profiles of individual differences in long-term adjustment to loss, according to psychological and biological markers over time; and 2) to examine whether cumulative lifetime stress exposure and neuro-inflammatory sensitivity to stress moderate the association between an acute stressful life event (i.e., the loss of a terminally-ill spouse after a long period of intensive caregiving) and the spouse's health outcomes following bereavement and, thereby, explain individual differences in resilience.

ELIGIBILITY:
Inclusion Criteria:

* Participant age ≥ 18 years
* Caregiver or spouse of a patients suffering from a terminal illness (estimated life expectancy ≤ 6 months),
* regarded as the patients primary caregiver (i.e., intimately involved in care of the patient since time of the diagnosis, looking after his/her daily needs, supervising the medications, bringing the patient to the hospital, staying with the patient during inpatient stay, and maintaining liaison with the hospital staff),
* German as primary language
* signed informed consent.

Exclusion Criteria:

* Significant visual or auditory problems, cognitive impairment,
* morbid obesity (body mass index ≥40 kg/m2,
* alcohol or drug abuse
* active malignancy
* severe illness (respiratory, heart, liver and renal failure)
* major medical conditions involving the immune system (e.g., diabetes type 1 or 2, autoimmune and/ or inflammatory diseases including rheumatoid arthritis and ulcerative colitis, asthma, thyroid diseases)
* severe hypertension (>200/120 mmHg)
* regular use of medication with major immunological consequences (e.g., corticosteroids, immunosuppressive therapy)
* pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Spouses or caregivers (N = 100) of patients suffering from an advanced cancer that is unlikely to be cured or controlled with treatment and is likely to cause death (estimated life expectancy of ≤ 6 months). Spouses/caregivers of severely ill cancer patients will be assigned to the study and followed for a period of one year. In addition, fifty gender and age-matched non-bereaved subjects will be recruited in the community. However, this control group will undergo only one assessment.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The Center for Epidemiological Studies Depression Scale (CES-D) | Assessment 1: 6 months before patient's death; Assessment: 3-6 months post-loss; Assessment: 9-12 months post-loss
  Depression
interleukine-6 (IL-6) | Assessment 1: 6 months before patient's death; Assessment: 3-6 months post-loss; Assessment: 9-12 months post-loss
  Measure of inflammation

SECONDARY OUTCOMES:
The Stress and Adversity Inventory (STRAIN) | Assessment 1: 6 months before patient's death
  Adverse life experiences
Physical Health Questionnaire (PHQ-D) | Assessment 1: 6 months before patient's death; Assessment: 3-6 months post-loss; Assessment: 9-12 months post-loss
  Physical Health
Charlson Comorbidity Index (CC) | Assessment 1: 6 months before patient's death; Assessment: 3-6 months post-loss; Assessment: 9-12 months post-loss
  Comorbidities
The Perceived Stress Scale (PSS) | Assessment 1: 6 months before patient's death; Assessment: 3-6 months post-loss; Assessment: 9-12 months post-loss
  Stress
The RAND 12-Item Short Form Health Survey (SF-12) | Assessment 1: 6 months before patient's death; Assessment: 3-6 months post-loss; Assessment: 9-12 months post-loss
  Quality of Life
Pittsburg Sleep Quality Index (PSQI) | Assessment 1: 6 months before patient's death; Assessment: 3-6 months post-loss; Assessment: 9-12 months post-loss
  Sleep quality
PTSD Checklist for DSM-5 (PCL-5) | Assessment 1: 6 months before patient's death; Assessment: 3-6 months post-loss; Assessment: 9-12 months post-loss
  PTSD symptoms
Dissociative Subtype of PTSD Scale (DSPS) | Assessment 1: 6 months before patient's death; Assessment: 3-6 months post-loss; Assessment: 9-12 months post-loss
  Dissociative symptomes
Cognitive Processing Questionnaire (CPQ) | Assessment 1: 6 months before patient's death; Assessment: 3-6 months post-loss; Assessment: 9-12 months post-loss
  Cognitive Processing
The Inventory of Complicated Grief (ICG) | Assessment 1: 6 months before patient's death; Assessment: 3-6 months post-loss; Assessment: 9-12 months post-loss
  Complicated grief
Prolonged Grief Reaction (PG13+9) | Assessment 1: 6 months before patient's death; Assessment: 3-6 months post-loss; Assessment: 9-12 months post-loss
  Prolonged grief
heart-rate/heart-rate variability | Assessment 1: 6 months before patient's death; Assessment: 3-6 months post-loss; Assessment: 9-12 months post-loss
  physiological stress marker
nail cortisol and cortisone | Assessment 1: 6 months before patient's death; Assessment: 3-6 months post-loss; Assessment: 9-12 months post-loss
  nail cortisol and cortisone
tumor necrosis factor alpha (TNF-a) | Assessment 1: 6 months before patient's death; Assessment: 3-6 months post-loss; Assessment: 9-12 months post-loss
  measure of inflammation
C-reactive protein (CRP) | Assessment 1: 6 months before patient's death; Assessment: 3-6 months post-loss; Assessment: 9-12 months post-loss
  measure of inflammation

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland